CLINICAL TRIAL: NCT02617563
Title: A Prospective, 5-Year Global Study on MAST™ Minimally Invasive Fusion Procedures for the Treatment of the Degenerative Lumbar Spine
Brief Title: 5-Year Global Study on MAST™ Minimally Invasive Fusion Procedures to Treat Degenerative Lumbar Spine (MASTERS-D2)
Acronym: MASTERS-D2
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-01
Record Dates: First submitted 2015-11-17; First posted 2015-12-01 (Estimated); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Intervertebral Disc Degeneration
Keywords: spondylolisthesis; CD Horizon® Spinal Systems; minimal invasive; Spinal Fusion; MAST procedure; Lumbar fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Minimally invasive lumbar fusion: A single or double level instrumented fusion using minimally invasive PLIF, TLIF, MIDLF, DLIF, OLIF, ALIF procedures for the treatment of the degenerative lumbar spine.
  Interventions: Device: Minimally invasive lumbar fusion

INTERVENTIONS:
Device: Minimally invasive lumbar fusion — Patients will receive a single or double level instrumented fusion using a minimally invasive/MAST™ PLIF, TLIF, DLIF, OLIF, ALIF or MIDLF surgical procedure with a posterior fixation. For the use of a posterior fixation system, the CD Horizon™ Spinal System, is mandatory in this study and will be either mini-open and/or percutaneous.

SUMMARY:
The purpose of this study is

* to evaluate the effectiveness of MAST techniques for anterior/lateral and posterior approaches in Degenerative Disc Disease (DDD) patients with spondylolisthesis (≥ grade I).
* To assess how single or double level MAST(Minimal Access Spinal Technologies) fusion procedures PLIF (Posterior Lumbar Interbody Fusion), TLIF (Transforaminal Lumbar Interbody Fusion), DLIF (Direct Lateral Interbody Fusion), OLIF (Oblique Lumbar Interbody Fusion), ALIF (Anterior Lumbar Interbody Fusion), or MIDLF (Midline Lumbar Interbody Fusion) are used in surgical practice and to describe long-term safety and effectiveness in a broad patient population of patients with degenerative lumbar disc disease .

DETAILED DESCRIPTION:
In this Prospective, Global (multi center), Post Market Release (PMR) Study, Patients will be submitted to a single or double level instrumented fusion procedure using a PLIF, TLIF, ALIF, OLIF, DLIF or MIDLF technique via a minimally invasive procedure and will receive the same medical treatment as if they would not participate in this study.

* The study will be monitored with visits conducted at the start, during and at the closure of the clinical study.
* MedDRA coding will be used to classify the Adverse Event.
* The study will be conducted according to Medtronic SOPs
* Sample size calculation: Assuming that the standard deviation for ODI improvement at 3 months is 20 for both groups (anterolateral and posterior) and there is no difference in the mean ODI improvement at 3 months, with 80% power and 5% alpha level, the sample size for the primary endpoint (DDD patients operated for spondylolisthesis) is as follows in order to claim equivalence between two groups with equivalent margin (-10, 10):
* Estimated sample size per group (anterolateral procedures versus posterior procedures): 70
* Estimated total sample size for spondylolisthesis patients: 140
* From the MASTERS-D study it is know that approximately 50% of the patients with degenerative disc disease have spondylolisthesis ≥ grade I. Hence the required total sample size is 140/0.5 = 280. The study is anticipated to enroll 350 patients.
* In addition to a final statistical analysis, 3 months and annual interim analyses are anticipated.
* The study hypothesis for the primary objective is to verify whether patients operated for spondylolisthesis (≥ grade I) have equivalent mean improvement of ODI at 3 months regardless of the minimally invasive surgical procedure (anterolateral or posterior) used.
* The null-hypothesis: Ho: Δ ODI_Anterolateral ≠ Δ ODI_posterior
* will be tested against the alternative hypothesis: HA: Δ ODI_Anterolateral = Δ ODI_posterior Where Δ ODI_Anterolateral is the average improvement in ODI score (baseline - 3 months) in spondylolisthesis subjects treated with the anterolateral approach and Δ ODI_posterior is the average improvement in ODI score (baseline - 3 months) in spondylolisthesis subjects treated with the posterior approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age (or minimum age as required by local regulations)
* Patient has degenerative disc disease and an indication for a single or double level instrumented lumbar fusion for the treatment
* Patient agrees to participate in the study and is able to sign the Data Release Form/Informed Consent
* The procedure planned for the patient complies with the labeling of the Devices that may be used in the surgical procedure as described in the section Medical Devices of the Clinical Investigation Plan
* Patient is planned to be submitted to a minimally invasive fusion procedure using a posterior (PLIF, TLIF, MIDLF) or anterolateral (OLIF, ALIF, DLIF ) technique*

  *For a double level instrumented fusion, the same procedure must be used for both levels.
* The patient is willing and is able to perform study procedures and required follow-up visits.

Exclusion Criteria:

* Patient that has already undergone a lumbar fusion surgery
* Patient that has already undergone open lumbar surgery other than standard decompression surgery
* Indications for the procedure other than degenerative spine disease like: Osteoporotic vertebral fractures, Spine trauma fractures or Spine tumor
* Illiterate or vulnerable patients (e.g. minors, participants incapable of judgment or participants under tutelage)
* Concurrent participation in another clinical study that may confound study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 361 patients suffering from lumbar degenerative disc disease (DDD) were enrolled over a period of 42 months in 27 sites located in Europe, Latin America, and Asia Pacific.
Sampling Method: Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2015-12; Primary Completion 2019-11-10 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Kepler Universitatsklinikum, Linz, Austria
- AZ Delta, Roeselare, Belgium
- Hospital Universitario Cajuru, Curitiba, Brazil
- China (3):
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Shangai Tenth People's Hospital, Shanghai
- Nový Hradec Králové, Hradec Králové, Czechia
- Glostrup Hospital, Glostrup Municipality, Denmark
- France (3):
  - Hôpital Civil de Strasbourg (NHC), Eckbolsheim
  - CHRU de Lille, Hôpital Roger Salengro, Lille
  - Service de Neurochirurgie la Timone, Marseille
- Klinikum Magdeburg, Magdeburg, Germany
- A.O. Fatebenefratelli e Oftalmico, Milan, Italy
- Hospital Naval General de Alta Especialidad, Mexico City, Mexico
- Portugal (2):
  - Hospital Escala Braga, Braga
  - Centro Hospitalar de Sao Joao, Porto
- Russia (2):
  - Nizhny Novgorod Research Institute of Traumatology and Orthopedics of Public Health Ministry, Nizhny Novgorod
  - Scientific Research Institute of Traumatology and Orthopedics, Novosibirsk
- A-klinik, Bratislava, Slovakia
- South Korea (3):
  - Department of Orthopedics, Korea University Ansan Hospital, Ansan
  - National Health Insurance Corporation Ilsan Hospital, Gyeonggi-do
  - Department of Neurological Surgery, Chung-Ang University Hospital, Seoul
- Spain (2):
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital L'Horta Manises, Valencia
- United Kingdom (2):
  - Hull Royal Infirmary, Hull
  - East Suffolk and North Essex NHS Foundation Trust (was formerly Ipswich Hospital NHS), Ipswich

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 361 patient enrolled, twenty-four participants were excluded after pre-op. The reasons for these exclusions were that these 24 participants did not undergo the minimally invasive fusion treatment per CIP
Groups:
- Total Population ANT: Participants who received anterolateral MI lumbar surgery (ALIF, DLIF or OLIF) with posterior fixation
- Total Population POST: Participants who received posterior MI lumbar surgery (MIDLF, PLIF or TLIF) with posterior fixation
Period: 4 Weeks
Arm/Group | Total Population ANT | Total Population POST
Started | 164 | 173
Completed | 162 | 173
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: 3 Months
Arm/Group | Total Population ANT | Total Population POST
Started | 162 | 173
Completed | 161 | 172
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: 1 Year
Arm/Group | Total Population ANT | Total Population POST
Started | 161 | 172
Completed | 160 | 170
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Period: 2 Year
Arm/Group | Total Population ANT | Total Population POST
Started | 160 | 170
Completed | 157 | 165
Not Completed | 3 | 5
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 4
Period: 3 Year
Arm/Group | Total Population ANT | Total Population POST
Started | 157 | 165
Completed | 153 | 160
Not Completed | 4 | 5
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Period: 4 Year
Arm/Group | Total Population ANT | Total Population POST
Started | 153 | 160
Completed | 146 | 158
Not Completed | 7 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1
Period: 5 Year
Arm/Group | Total Population ANT | Total Population POST
Started | 146 | 158
Completed | 136 | 152
Not Completed | 10 | 6
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 9 | 5
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Population ANT | Total Population POST | Total
Number analyzed (Participants) | 164 | 173 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.3) | 59.7 (11.1) | 58.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 103 | 203
  Male | 64 | 70 | 134
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Argentina | 3 | 3 | 6
  Czechia | 0 | 13 | 13
  United Kingdom | 11 | 17 | 28
  Portugal | 17 | 22 | 39
  Spain | 39 | 2 | 41
  Russia | 22 | 12 | 34
  South Korea | 26 | 23 | 49
  Austria | 9 | 5 | 14
  Belgium | 0 | 8 | 8
  China | 0 | 48 | 48
  Denmark | 1 | 1 | 2
  Brazil | 7 | 3 | 10
  Italy | 1 | 1 | 2
  Mexico | 0 | 1 | 1
  Slovakia | 0 | 3 | 3
  France | 28 | 7 | 35
  Germany | 0 | 4 | 4
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: One (1) patient didn't enter data on height, therefore BMI couldn't be calculated for this patient
  kg/m^2
    number analyzed (Participants) | 163 | 173 | 336
    (all) | 27.7 (4.9) | 26.8 (4.5) | 27.2 (4.7)
Current tobacco use [Count of Participants; unit: Participants]
  Uses tobacco | 38 | 33 | 71
  Does not use tobacco | 126 | 140 | 266
Working status [Count of Participants; unit: Participants]
  Not employed | 91 | 119 | 210
  Employed or independent worker | 73 | 54 | 127
History of spine surgery [Count of Participants; unit: Participants]
  Yes | 20 | 15 | 35
  No | 144 | 158 | 302
Medication use at baseline (Nonopioid) [Count of Participants; unit: Participants]
  Yes | 121 | 101 | 222
  No | 43 | 72 | 115
Medication use at baseline (Opioid) [Count of Participants; unit: Participants]
  Yes | 70 | 49 | 119
  No | 94 | 124 | 218
Medication use at baseline (Other) [Count of Participants; unit: Participants]
  Yes | 83 | 37 | 120
  No | 81 | 136 | 217

OUTCOME MEASURES:

1. Primary Outcome: Change (Preop-postop) of Disability, Oswestry Disability Index (ODI) at 3 Months as Compared to Baseline in DDD Patients With Spondylolisthesis
Description: To demonstrate that DDD patients operated for spondylolisthesis fare equally well regardless of the surgical procedure (anterolateral or posterior) performed as measured by the change of ODI at 3 months as compared to baseline.
  ODI=Oswestry Disability Scale [0-100]; higher scores mean a worse outcome Timepoints: Baseline and 3 months
Time Frame: 3 months
Population: 227 participants with spondylolisthesis were categorized into either ANT or POST groups, depending on the type of MI lumbar surgery received. n=206 of these patients completed the 3-month follow-up visit.
Measure: Mean (Standard Deviation); unit: change of score on a scale (ODI)
Groups:
- Spondylolisthesis ANT: Participants with spondylolisthesis who received anterolateral MI lumbar surgery (ALIF, DLIF or OLIF)
- Spondylolisthesis POST: Participants with spondylolisthesis who received posterior MI lumbar surgery (MIDLF, PLIF or TLIF)
Arm/Group | Spondylolisthesis ANT | Spondylolisthesis POST
Number analyzed (Participants) | 106 | 100
change of score on a scale (ODI) | 23.19 (21.32) | 26.08 (19.47)
Statistical Analysis 1: Comparison: Spondylolisthesis ANT vs Spondylolisthesis POST; Test type: Equivalence — ANCOVA was performed with baseline ODI as covariate, and two-sided 95% confidence interval (CI) for the least square mean difference of ODI improvement between two groups was calculated to test the hypothesis for the primary objective; p = 0.426, ANCOVA; Difference of Least Square Means = -1.76, 95% CI 2-sided [-6.11 to 2.59]

2. Secondary Outcome: Change (Preop-postop) in Disability ODI as Compared to Baseline in DDD Patients Without Spondylolisthesis
Description: To evaluate whether DDD patients without spondylolisthesis fare equally well regardless of the surgical procedure (anterolateral or posterior) performed, as measured by Oswestry Disability Index (ODI) at 3 months. Scored [0-100]; higher scores mean a worse outcome Timepoints: Baseline and 3 months
Time Frame: 3 months
Population: n=100 patients without spondylolisthesis completed the 3-month follow up, out of a total of n=110 non-spondilolisthesis patients enrolled
Measure: Mean (Standard Deviation); unit: score on a scale (improvement)
Groups:
- Non-spondylolisthesis ANT: Patients without spondylolisthesis who received anterolateral MI lumbar surgery (ALIF, DLIF or OLIF) with posterior fixation
- Non-spondylolisthesis POST: Patients without spondylolisthesis who received posterior MI lumbar surgery (MIDLF, PLIF, TLIF) with posterior fixation
Arm/Group | Non-spondylolisthesis ANT | Non-spondylolisthesis POST
Number analyzed (Participants) | 46 | 53
score on a scale (improvement) | 13.41 (22.09) | 24.20 (20.02)

3. Secondary Outcome: Change (Preop-postop) in ODI Scores for the Total Population
Description: To observe the change in ODI scores as compared to baseline through 5 years. The score at baseline gives the baseline score [0-100]; the higher the score, the worse the outcome. Additional scores are based on the change from baseline. The higher the score, the greater the improvement.
  Timepoints: Baseline, 4 weeks, 3 months, 1-,2-,3-,4-, and 5-years
Time Frame: Through 5 years
Population: Participant numbers may deviate per follow-up visit due to data not having been completed for a number of participants (e.g. data not completed by follow-up, drop-out)
Measure: Mean (Standard Deviation); unit: score on a scale (improvement)
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
score on a scale (improvement)
  Baseline (score): number analyzed (Participants) | 163 | 173
  Baseline (score) | 46.46 (18.05) | 47.02 (15.89)
  4 Weeks: number analyzed (Participants) | 150 | 148
  4 Weeks | 13.27 (22.56) | 17.57 (19.87)
  3 Months: number analyzed (Participants) | 152 | 153
  3 Months | 20.23 (21.95) | 25.43 (19.62)
  1 Year: number analyzed (Participants) | 150 | 151
  1 Year | 24.47 (22.30) | 29.42 (19.63)
  2 Year: number analyzed (Participants) | 140 | 152
  2 Year | 27.80 (23.81) | 30.31 (20.52)
  3 Year: number analyzed (Participants) | 138 | 149
  3 Year | 27.15 (23.93) | 29.83 (21.08)
  4 Year: number analyzed (Participants) | 132 | 146
  4 Year | 26.08 (25.48) | 27.30 (21.01)
  5 Year: number analyzed (Participants) | 135 | 145
  5 Year | 26.55 (25.50) | 29.26 (19.67)

4. Secondary Outcome: Change (Preop-postop) in Visual Analog Scale (VAS) Back Pain Intensity
Description: To observe a change in VAS back pain as compared to baseline through 5 years. At baseline scored on a scale from [0-10]; 0 = No pain 10= Worst pain possible.
  Timepoints: Baseline, 4 weeks, 3 months, 1-,2-,3-,4-, and 5-years
Time Frame: Through 5 years
Population: Participant numbers may differ at follow-up time points due to data not being available for some (e.g. participant did not complete the data, or drop-out)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
score on a scale
  Baseline (score): number analyzed (Participants) | 163 | 173
  Baseline (score) | 6.48 (2.33) | 5.76 (2.76)
  4 Weeks: number analyzed (Participants) | 149 | 149
  4 Weeks | 3.48 (3.15) | 3.06 (3.06)
  3 Months: number analyzed (Participants) | 153 | 153
  3 Months | 3.47 (3.11) | 3.25 (3.23)
  1 Year: number analyzed (Participants) | 150 | 151
  1 Year | 3.48 (3.36) | 3.46 (3.01)
  2 Year: number analyzed (Participants) | 141 | 151
  2 Year | 3.50 (3.40) | 3.59 (3.01)
  3 Year: number analyzed (Participants) | 138 | 149
  3 Year | 3.54 (3.26) | 3.54 (2.92)
  4 Year: number analyzed (Participants) | 131 | 146
  4 Year | 3.42 (3.39) | 3.33 (3.04)
  5 Year: number analyzed (Participants) | 134 | 145
  5 Year | 3.90 (3.25) | 3.48 (2.93)

5. Secondary Outcome: Change (Preop-postop) in VAS Leg Pain Intensity
Description: To observe the change in VAS leg pain as compared to baseline through 5 years. The score at baseline gives the baseline score [0-10]; 0 = No pain 10= Worst pain possible.
  Timepoints: Baseline, 4 weeks, 3 months, 1-,2-,3-,4-, and 5-years
Time Frame: Through 5 years
Population: Number of participants may differ as data is not always available for all (e.g. data not completed by participant, drop-out)
Measure: Mean (Standard Deviation); unit: score on a scale (improvement)
Groups:
- Total Population POST: Participants who received posterior MI lumbar surgery (MIDLF, PLIF and TLIF) with posterior fixation
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
score on a scale (improvement)
  Baseline (score): number analyzed (Participants) | 162 | 173
  Baseline (score) | 6.18 (2.70) | 6.33 (2.57)
  4 Weeks: number analyzed (Participants) | 149 | 149
  4 Weeks | 3.79 (3.58) | 4.64 (3.25)
  3 Months: number analyzed (Participants) | 152 | 153
  3 Months | 3.99 (3.56) | 4.76 (3.44)
  1 Year: number analyzed (Participants) | 149 | 151
  1 Year | 3.83 (3.70) | 4.50 (3.57)
  2 Year: number analyzed (Participants) | 140 | 151
  2 Year | 4.17 (3.81) | 4.84 (3.49)
  3 Year: number analyzed (Participants) | 137 | 149
  3 Year | 4.18 (3.73) | 4.62 (3.51)
  4 Year: number analyzed (Participants) | 130 | 146
  4 Year | 3.58 (4.10) | 4.52 (3.50)
  5 Year: number analyzed (Participants) | 133 | 145
  5 Year | 4.23 (3.69) | 4.65 (3.40)

6. Secondary Outcome: Change (Postop-preop) in EQ-5D Index Score
Description: To observe the change in EuroQol-5 Dimension (EQ-5D) index score as compared to baseline through 5 years. Scored from [-0.109 to 1]. A higher score means a better outcome.
  Timepoints: Baseline, 4 weeks, 3 months, 1-,2-,3-,4-, and 5-years
Time Frame: Through 5 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale (improvement)
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
score on a scale (improvement)
  Baseline (score): number analyzed (Participants) | 159 | 172
  Baseline (score) | 0.492 (0.225) | 0.543 (0.226)
  4 Weeks: number analyzed (Participants) | 147 | 146
  4 Weeks | 0.209 (0.271) | 0.237 (0.246)
  3 Months: number analyzed (Participants) | 149 | 151
  3 Months | 0.267 (0.268) | 0.285 (0.248)
  1 Year: number analyzed (Participants) | 146 | 151
  1 Year | 0.261 (0.283) | 0.287 (0.239)
  2 Year: number analyzed (Participants) | 137 | 151
  2 Year | 0.307 (0.286) | 0.314 (0.257)
  3 Year: number analyzed (Participants) | 135 | 148
  3 Year | 0.301 (0.291) | 0.315 (0.247)
  4 Year: number analyzed (Participants) | 128 | 145
  4 Year | 0.284 (0.316) | 0.286 (0.249)
  5 Year: number analyzed (Participants) | 129 | 143
  5 Year | 0.300 (0.306) | 0.291 (0.249)

7. Secondary Outcome: The Neurological Success Rate
Description: Neurological status is based on four types of measurements (sections): motor, sensory, reflexes, and straight leg raising.
  Overall neurological success is defined as maintenance or improvement in all sections (motor, sensory, reflex, and straight leg raising) for the time period evaluated. In order for a section to be considered a success, each element in the section must remain the same or improve from the time of the baseline evaluation to the time period evaluated. Therefore, if any one element in any section does not stay the same or improve, then a patient was not considered a success for neurological status.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 54 | 59
Participants
  Motor function: Normal | 52 | 58
  Motor function: Abnormal | 2 | 1
  Sensory function: Normal | 53 | 57
  Sensory function: Abnormal | 1 | 2
  Reflexes: Normal | 54 | 58
  Reflexes: Abnormal | 0 | 1
  Straight leg raise: Normal | 53 | 59
  Straight leg raise: Abnormal | 1 | 0
  Overall Neurological Status: Normal | 51 | 56
  Overall Neurological Status: Abnormal | 3 | 3

8. Secondary Outcome: Fusion Success
Description: Fusion success rate was summarized for at 1, 2, 3, 4, 5 year follow-up. If a participant showed fusion success at early time points and non-fusion at a later time point, the fusion status at all earlier points was considered as non-fusion. For 2-level fusion participants, fusion success was defined as achieving fusion at both treated levels.
Time Frame: Through 5 years
Population: Fusion assessments weren't conducted at each time point for each participant, and not all participants had their fusion status assessed, hence the participant numbers are different at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
Participants
  12 Months: number analyzed (Participants) | 127 | 116
  12 Months: Fused | 110 | 100
  12 Months: Not Fused | 17 | 16
  24 Months: number analyzed (Participants) | 35 | 28
  24 Months: Fused | 33 | 25
  24 Months: Not Fused | 2 | 3
  36 Months: number analyzed (Participants) | 20 | 21
  36 Months: Fused | 19 | 18
  36 Months: Not Fused | 1 | 3
  48 Months: number analyzed (Participants) | 14 | 20
  48 Months: Fused | 13 | 20
  48 Months: Not Fused | 1 | 0
  60 Months: number analyzed (Participants) | 13 | 18
  60 Months: Fused | 12 | 18
  60 Months: Not Fused | 1 | 0
  The Last Evaluation of Fusion Status: number analyzed (Participants) | 143 | 130
  The Last Evaluation of Fusion Status: Fused | 127 | 115
  The Last Evaluation of Fusion Status: Not Fused | 16 | 15

9. Secondary Outcome: Proportion of Patients Needing a Secondary Spinal Surgery at the Index and/or Adjacent Level(s) (Reoperation Rates) Throughout the Study
Description: To document Secondary Surgeries at index and/or adjacent level(s)throughout the study. When a participant requires additional surgery at the index level(s), it can be an indicator of insufficient outcomes of the initial surgery. Due to the progressive nature of the degenerative lumbar spine, additional surgeries at the index and/or adjacent levels might be required after the initial surgery. To ensure all safety and economic values are collected, the revision surgeries and their complication types and rates will be assessed during the study by the surgeons.
  For secondary surgery at index levels and/or secondary surgery at adjacent levels, survival analysis was performed to estimate the cumulative event rate up to 5 years.
Time Frame: Through 5 years
Population: Not all participants had additional surgery, and some participants had multiple revision surgeries. In the ANT group n=16 participants who had at least 1 revision surgery, in the POST group n=21.
Measure: Number; unit: number of revision surgeries
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
number of revision surgeries
  Index levels only | 6 | 13
  Adjacent levels only | 4 | 8
  Both index and adjacent levels | 2 | 2
  Others | 6 | 1

10. Secondary Outcome: Adverse Events
Description: Document Adverse Events occurrence throughout the study
Time Frame: Through 5 years
Measure: Number; unit: Adverse Events (n)
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
Adverse Events (n)
  Device-related | 10 | 5
  MAST/MI (minimally invasive)-related | 18 | 17
  General Surgery-related | 66 | 75
  Disease-related | 63 | 61

11. Secondary Outcome: Amount of Days Needed for First Ambulation
Description: To observe and document the days needed for participants to get out of bed and ambulate with or without assistance. Time range: [0-11] days
Time Frame: From surgery up to hospital discharge, up to 11 days
Population: For two participants in the ANT arm, no data was available for "Time needed for first ambulation"
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 162 | 173
Days | 1.6 (1.3) | 1.9 (1.6)

12. Secondary Outcome: Amount of Days Needed to Recover From Surgery
Description: To observe and document the days after the surgery, fulfilling following criteria:
  * No need for intravenous infusion of analgesic drugs
  * No ongoing surgery related adverse events impending discharge
  * No need for nursing care
  Timeframe: [0-46] days
  The objective of the Surgery Recovery Day assessment is to collect the day when the participant could be discharged based on his actual clinical condition because the effective day of discharge may be prolonged by factors other than the participant's clinical recovery such as social factors or co-morbidity.
  For the purpose of reporting these parameters the day of the surgery were considered 'D0', the first day after surgery as 'D1', the second day as 'D2' and so on.
Time Frame: Surgery Recovery Day up to hospital discharge, with a maximum of 46 days
Population: Data for 1 participant in the ANT group is unavailable for "Surgery Recovery"
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 163 | 173
Days | 4.4 (3.7) | 5.0 (5.2)

13. Secondary Outcome: Healthcare Economics Evaluation "Medications"
Description: Healthcare utilization were measured with the following three costs components:
  1. resources: surgery room, length of hospital stay, additional medical visits (outpatient consultations, visits to primary care services, etc)
  2. medications
  3. non-pharmacologic therapies: rehabilitation program
Time Frame: Baseline to 5-year follow-up
Population: Not all data completed for each participant at each follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
Participants
  Baseline : Nonopioid analgesics: Yes | 121 | 101
  Baseline : Nonopioid analgesics: No | 43 | 72
  Baseline : Opioid analgesics: Yes | 70 | 49
  Baseline : Opioid analgesics: No | 94 | 124
  Baseline : Other medications: Yes | 83 | 37
  Baseline : Other medications: No | 81 | 136
  4 Weeks : Nonopioid analgesics: number analyzed (Participants) | 154 | 157
  4 Weeks : Nonopioid analgesics: Yes | 99 | 89
  4 Weeks : Nonopioid analgesics: No | 55 | 68
  4 Weeks : Opioid analgesics: number analyzed (Participants) | 154 | 157
  4 Weeks : Opioid analgesics: Yes | 53 | 42
  4 Weeks : Opioid analgesics: No | 101 | 115
  4 Weeks : Other medications: number analyzed (Participants) | 154 | 157
  4 Weeks : Other medications: Yes | 75 | 32
  4 Weeks : Other medications: No | 79 | 125
  3 Months : Nonopioid analgesics: number analyzed (Participants) | 159 | 160
  3 Months : Nonopioid analgesics: Yes | 97 | 68
  3 Months : Nonopioid analgesics: No | 62 | 92
  3 Months : Opioid analgesics: number analyzed (Participants) | 159 | 160
  3 Months : Opioid analgesics: Yes | 48 | 29
  3 Months : Opioid analgesics: No | 111 | 131
  3 Months : Other medications: number analyzed (Participants) | 159 | 160
  3 Months : Other medications: Yes | 67 | 23
  3 Months : Other medications: No | 92 | 137
  1 Year : Nonopioid analgesics: number analyzed (Participants) | 152 | 158
  1 Year : Nonopioid analgesics: Yes | 73 | 53
  1 Year : Nonopioid analgesics: No | 79 | 105
  1 Year : Opioid analgesics: number analyzed (Participants) | 152 | 158
  1 Year : Opioid analgesics: Yes | 29 | 16
  1 Year : Opioid analgesics: No | 123 | 142
  1 Year : Other medications: number analyzed (Participants) | 152 | 158
  1 Year : Other medications: Yes | 55 | 24
  1 Year : Other medications: No | 97 | 134
  2 Year : Nonopioid analgesics: number analyzed (Participants) | 147 | 157
  2 Year : Nonopioid analgesics: Yes | 56 | 48
  2 Year : Nonopioid analgesics: No | 91 | 109
  2 Year : Opioid analgesics: number analyzed (Participants) | 147 | 157
  2 Year : Opioid analgesics: Yes | 24 | 16
  2 Year : Opioid analgesics: No | 123 | 141
  2 Year : Other medications: number analyzed (Participants) | 147 | 157
  2 Year : Other medications: Yes | 50 | 27
  2 Year : Other medications: No | 97 | 130
  3 Year : Nonopioid analgesics: number analyzed (Participants) | 144 | 154
  3 Year : Nonopioid analgesics: Yes | 57 | 48
  3 Year : Nonopioid analgesics: No | 87 | 106
  3 Year : Opioid analgesics: number analyzed (Participants) | 144 | 154
  3 Year : Opioid analgesics: Yes | 18 | 8
  3 Year : Opioid analgesics: No | 126 | 146
  3 Year : Other medications: number analyzed (Participants) | 144 | 154
  3 Year : Other medications: Yes | 46 | 23
  3 Year : Other medications: No | 98 | 131
  4 Year : Nonopioid analgesics: number analyzed (Participants) | 133 | 152
  4 Year : Nonopioid analgesics: Yes | 44 | 45
  4 Year : Nonopioid analgesics: No | 89 | 107
  4 Year : Opioid analgesics: number analyzed (Participants) | 133 | 152
  4 Year : Opioid analgesics: Yes | 21 | 10
  4 Year : Opioid analgesics: No | 112 | 142
  4 Year : Other medications: number analyzed (Participants) | 133 | 152
  4 Year : Other medications: Yes | 38 | 26
  4 Year : Other medications: No | 95 | 126
  5 Year : Nonopioid analgesics: number analyzed (Participants) | 135 | 151
  5 Year : Nonopioid analgesics: Yes | 38 | 41
  5 Year : Nonopioid analgesics: No | 97 | 110
  5 Year : Opioid analgesics: number analyzed (Participants) | 135 | 151
  5 Year : Opioid analgesics: Yes | 20 | 10
  5 Year : Opioid analgesics: No | 115 | 141
  5 Year : Other medications: number analyzed (Participants) | 135 | 151
  5 Year : Other medications: Yes | 34 | 29
  5 Year : Other medications: No | 101 | 122

14. Secondary Outcome: Health Economics Evaluation "Resources"
Description: Healthcare utilization is measured with the following three cost components:
  1. resources: surgery room, length of hospital stay, additional medical visits (outpatient consultations, visits to primary care services, etc)
  2. medications
  3. non-pharmacologic therapies: rehabilitation program
Time Frame: Through 5 years
Population: Some questions were left blank by the sites.
Measure: Mean (Standard Deviation); unit: Number of occurrences
Groups:
- Total Study Population ANT: Participants who received anterolateral MI lumbar surgery (ALIF, DLIF, OLIF) with posterior fixation
- Total Study Population POST: Participants who received posterior MI lumbar surgery (MIDLF, PLIF, TLIF) with posterior fixation
Arm/Group | Total Study Population ANT | Total Study Population POST
Number analyzed (Participants) | 164 | 173
Number of occurrences
  Nr of times patient received care in outpatient centre due to back pain at 5 years: number analyzed (Participants) | 6 | 5
  Nr of times patient received care in outpatient centre due to back pain at 5 years | 2.2 (1.6) | 3.6 (3.6)
  Nr of times patient received care in primary care service due to back pain at 5 years: number analyzed (Participants) | 4 | 11
  Nr of times patient received care in primary care service due to back pain at 5 years | 1.8 (0.5) | 2.2 (1.1)

15. Secondary Outcome: Health Economics Evaluation "Rehabilitation Program"
Description: Healthcare utilization is measured with the following three costs components:
  1. resources: surgery room, length of hospital stay, additional medical visits (outpatient consultations, visits to primary care services, etc)
  2. medications
  3. non-pharmacologic therapies: rehabilitation program
Time Frame: Baseline to 5 years
Population: Data was not always completed for each participant by the site
Measure: Count of Participants; unit: Participants
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 164 | 173
Participants
  Discharge :Will the patient be transferred to a Rehabilitation center?: number analyzed (Participants) | 163 | 173
  Discharge :Will the patient be transferred to a Rehabilitation center?: Yes | 9 | 6
  Discharge :Will the patient be transferred to a Rehabilitation center?: No | 154 | 167
  Discharge : Rehabilitation care at home: number analyzed (Participants) | 163 | 173
  Discharge : Rehabilitation care at home: Yes | 22 | 21
  Discharge : Rehabilitation care at home: No | 141 | 152
  Discharge : Care at an outpatient rehabilitation center: number analyzed (Participants) | 163 | 173
  Discharge : Care at an outpatient rehabilitation center: Yes | 15 | 42
  Discharge : Care at an outpatient rehabilitation center: No | 148 | 131
  4 Weeks: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: number analyzed (Participants) | 154 | 157
  4 Weeks: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: Yes | 20 | 8
  4 Weeks: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: No | 134 | 149
  4 Weeks : Rehab center: number analyzed (Participants) | 19 | 8
  4 Weeks : Rehab center: Yes | 4 | 3
  4 Weeks : Rehab center: No | 15 | 5
  4 Weeks : Rehabilitation care at home: number analyzed (Participants) | 19 | 8
  4 Weeks : Rehabilitation care at home: Yes | 11 | 1
  4 Weeks : Rehabilitation care at home: No | 8 | 7
  4 Weeks : Care at an outpatient rehabilitation center: number analyzed (Participants) | 19 | 8
  4 Weeks : Care at an outpatient rehabilitation center: Yes | 5 | 5
  4 Weeks : Care at an outpatient rehabilitation center: No | 14 | 3
  3 Months: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: number analyzed (Participants) | 159 | 160
  3 Months: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: Yes | 34 | 36
  3 Months: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: No | 125 | 124
  3 Months : Rehab center: number analyzed (Participants) | 34 | 36
  3 Months : Rehab center: Yes | 6 | 9
  3 Months : Rehab center: No | 28 | 27
  3 Months : Rehabilitation care at home: number analyzed (Participants) | 34 | 36
  3 Months : Rehabilitation care at home: Yes | 3 | 6
  3 Months : Rehabilitation care at home: No | 31 | 30
  3 Months : Care at an outpatient rehabilitation center: number analyzed (Participants) | 34 | 36
  3 Months : Care at an outpatient rehabilitation center: Yes | 27 | 22
  3 Months : Care at an outpatient rehabilitation center: No | 7 | 14
  1 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: number analyzed (Participants) | 152 | 158
  1 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: Yes | 27 | 27
  1 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: No | 125 | 131
  1 Year : Rehab center: number analyzed (Participants) | 27 | 26
  1 Year : Rehab center: Yes | 12 | 8
  1 Year : Rehab center: No | 15 | 18
  1 Year : Rehabilitation care at home: number analyzed (Participants) | 27 | 26
  1 Year : Rehabilitation care at home: Yes | 2 | 1
  1 Year : Rehabilitation care at home: No | 25 | 25
  1 Year : Care at an outpatient rehabilitation center: number analyzed (Participants) | 27 | 26
  1 Year : Care at an outpatient rehabilitation center: Yes | 22 | 18
  1 Year : Care at an outpatient rehabilitation center: No | 5 | 8
  2 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: number analyzed (Participants) | 147 | 157
  2 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: Yes | 9 | 9
  2 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: No | 138 | 148
  2 Year : Rehab center: number analyzed (Participants) | 9 | 9
  2 Year : Rehab center: Yes | 1 | 2
  2 Year : Rehab center: No | 8 | 7
  2 Year : Rehabilitation care at home: number analyzed (Participants) | 9 | 9
  2 Year : Rehabilitation care at home: Yes | 1 | 0
  2 Year : Rehabilitation care at home: No | 8 | 9
  2 Year : Care at an outpatient rehabilitation center: number analyzed (Participants) | 9 | 9
  2 Year : Care at an outpatient rehabilitation center: Yes | 7 | 7
  2 Year : Care at an outpatient rehabilitation center: No | 2 | 2
  3 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: number analyzed (Participants) | 145 | 154
  3 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: Yes | 6 | 9
  3 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: No | 139 | 145
  3 Year : Rehab center: number analyzed (Participants) | 6 | 8
  3 Year : Rehab center: Yes | 2 | 3
  3 Year : Rehab center: No | 4 | 5
  3 Year : Rehabilitation care at home: number analyzed (Participants) | 6 | 8
  3 Year : Rehabilitation care at home: Yes | 2 | 0
  3 Year : Rehabilitation care at home: No | 4 | 8
  3 Year : Care at an outpatient rehabilitation center: number analyzed (Participants) | 6 | 8
  3 Year : Care at an outpatient rehabilitation center: Yes | 2 | 5
  3 Year : Care at an outpatient rehabilitation center: No | 4 | 3
  4 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: number analyzed (Participants) | 133 | 152
  4 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: Yes | 3 | 10
  4 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: No | 130 | 142
  4 Year : Rehab center: number analyzed (Participants) | 3 | 10
  4 Year : Rehab center: Yes | 0 | 3
  4 Year : Rehab center: No | 3 | 7
  4 Year : Rehabilitation care at home: number analyzed (Participants) | 3 | 10
  4 Year : Rehabilitation care at home: Yes | 0 | 1
  4 Year : Rehabilitation care at home: No | 3 | 9
  4 Year : Care at an outpatient rehabilitation center: number analyzed (Participants) | 3 | 10
  4 Year : Care at an outpatient rehabilitation center: Yes | 3 | 6
  4 Year : Care at an outpatient rehabilitation center: No | 0 | 4
  5 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: number analyzed (Participants) | 135 | 151
  5 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: Yes | 4 | 3
  5 Year: Any Rehabilitation Program Between This Scheduled Visit and the Previous Scheduled Visit: No | 131 | 148
  5 Year : Rehab center: number analyzed (Participants) | 4 | 3
  5 Year : Rehab center: Yes | 1 | 1
  5 Year : Rehab center: No | 3 | 2
  5 Year : Rehabilitation care at home: number analyzed (Participants) | 4 | 3
  5 Year : Rehabilitation care at home: Yes | 0 | 1
  5 Year : Rehabilitation care at home: No | 4 | 2
  5 Year : Care at an outpatient rehabilitation center: number analyzed (Participants) | 4 | 3
  5 Year : Care at an outpatient rehabilitation center: Yes | 3 | 1
  5 Year : Care at an outpatient rehabilitation center: No | 1 | 2

16. Secondary Outcome: Health Economics Evaluation "Operative Time"
Description: as for outcome 14
Time Frame: Peri-operative
Population: Some questions were left blank by the sites
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 162 | 171
hours | 3.371 (1.279) | 2.860 (1.028)

17. Secondary Outcome: Health Economics Evaluation "Estimated Blood Loss"
Description: as for outcome 14
Time Frame: Peri-operative
Population: Some questions were left blank by the sites
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 155 | 166
ml | 148.2 (201.5) | 296.3 (238.7)

18. Secondary Outcome: Health Economics Evaluation "Length of Hospital Stay"
Description: Healthcare utilization is measured with the following three cost components:
  1. resources: surgery room, length of hospital stay, additional medical visits (outpatient consultations, visits to primary care services, etc)
  2. medications
  3. non-pharmacologic therapies: rehabilitation program
  The minimum-maximum time spent at the hospital was [1-53 days]
Time Frame: Post-operative, up to 53 days
Population: Some questions were left blank by the sites
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 163 | 173
Days | 6.6 (5.4) | 7.5 (5.9)

19. Secondary Outcome: Health Economics Evaluation "Total Fluoroscopy Time"
Description: as for outcome 14
Time Frame: Peri-operative
Population: Some questions were left blank by the sites
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Total Population ANT | Total Population POST
Number analyzed (Participants) | 150 | 166
seconds | 144.8 (151.0) | 143.5 (202.9)

20. Secondary Outcome: To Observe and Document the Patient Profile When Choosing a Particular Minimally Invasive Fusion Procedure - Categorical Variables
Description: To observe and document the patient profile when choosing a particular minimally invasive fusion procedure:
  Baseline information is summarized for all DDD patients per surgical procedure (ALIF, OLIF, DLIF, PLIF, TLIF, MIDLF).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- ALIF: Patients who received ALIF MI lumbar surgery
- DLIF: Patients who received DLIF MI lumbar surgery
- OLIF: Patients who received OLIF MI lumbar surgery
- PLIF: Patients who received PLIF MI lumbar surgery
- MIDLF: Patients who received MIDLF MI lumbar surgery
- TLIF: Patients who received TLIF MI lumbar surgery
Arm/Group | ALIF | DLIF | OLIF | PLIF | MIDLF | TLIF
Number analyzed (Participants) | 43 | 50 | 71 | 22 | 65 | 86
Participants
  Gender: Female?: Yes | 20 | 27 | 53 | 11 | 43 | 49
  Gender: Female?: No | 23 | 23 | 18 | 11 | 22 | 37
  Does the patient currently use tobacco?: Yes | 18 | 10 | 10 | 6 | 6 | 21
  Does the patient currently use tobacco?: No | 25 | 40 | 61 | 16 | 59 | 65
  Preoperative work status: Employed/independent worker?: Yes | 27 | 22 | 24 | 9 | 23 | 22
  Preoperative work status: Employed/independent worker?: No | 16 | 28 | 47 | 13 | 42 | 64

21. Secondary Outcome: To Observe and Document the Patient Profile When Choosing a Particular Minimally Invasive Fusion Procedure - Age
Description: as for outcome 20
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: years
Groups:
- ALIF: Participants who received ALIF MI lumbar surgery
- DLIF: Participants who received DLIF MI lumbar surgery
- OLIF: Participants who received OLIF MI lumbar surgery
- PLIF: Participants who received PLIF MI lumbar surgery
- MIDLF: Participants who received MIDLF MI lumbar surgery
- TLIF: Participants who received TLIF MI lumbar surgery
Arm/Group | ALIF | DLIF | OLIF | PLIF | MIDLF | TLIF
Number analyzed (Participants) | 43 | 50 | 71 | 22 | 65 | 86
years | 49.4 (9.5) | 59.5 (9.0) | 60.5 (9.2) | 54.5 (10.8) | 61.3 (10.6) | 59.8 (11.3)

22. Secondary Outcome: To Observe and Document the Patient Profile When Choosing a Particular Minimally Invasive Fusion Procedure - Height
Description: as for outcome 20
Time Frame: Baseline
Population: For one participant in the OLIF Arm/Group height wasn't provided on the eCRF
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | ALIF | DLIF | OLIF | PLIF | MIDLF | TLIF
Number analyzed (Participants) | 43 | 50 | 70 | 22 | 65 | 86
centimeter (cm) | 169.4 (9.0) | 167.5 (9.6) | 162.3 (8.7) | 167.3 (8.1) | 164.0 (10.4) | 164.2 (8.2)

23. Secondary Outcome: To Observe and Document the Patient Profile When Choosing a Particular Minimally Invasive Fusion Procedure - Weight
Description: as for outcome 20
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | ALIF | DLIF | OLIF | PLIF | MIDLF | TLIF
Number analyzed (Participants) | 43 | 50 | 71 | 22 | 65 | 86
kilogram (kg) | 77.2 (15.2) | 82.3 (15.5) | 71.4 (13.8) | 80.9 (15.3) | 75.2 (18.6) | 69.4 (13.1)

24. Secondary Outcome: To Observe and Document the Patient Profile When Choosing a Particular Minimally Invasive Fusion Procedure - BMI
Description: as for outcome 20
Time Frame: Baseline
Population: For one participant height wasn't provided on the eCRF, hence this data and the BMI calculation are not available for this participant.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | ALIF | DLIF | OLIF | PLIF | MIDLF | TLIF
Number analyzed (Participants) | 43 | 50 | 70 | 22 | 65 | 86
kg/m2 | 26.8 (4.2) | 29.4 (5.6) | 27.0 (4.3) | 28.9 (5.0) | 27.7 (5.1) | 25.6 (3.5)

ADVERSE EVENTS:
Time Frame: The data was collected from Baseline until the 5-year follow-up visit.
Description: AE reporting through systematic assessment: at each follow-up visit site personnel was asked to review if new AEs had occurred since the previous visit.
  For the non-serious AE we have only reported those cases that occurred in 5% or more of the patients (at least in one arm), as is detailed below. The total number of patients who experienced any (i.e. including those that occurred in <5% and >=5% of the patients ) non-serious AE in the Anterolateral group is 114, and the Posterior group is 104.
Arm/Group | Total Population ANT | Total Population POST
All-Cause Mortality (participants affected / at risk) | 4/164 | 2/173
Serious Adverse Events (participants affected / at risk) | 58/164 | 55/173
Other Adverse Events (participants affected / at risk) | 56/164 | 43/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Population ANT (N=164) | Total Population POST (N=173)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial Fibrilation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Congenital foot malformation (Congenital, familial and genetic disorders) | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 4
Cataract nuclear (Eye disorders) | 0 | 1
Optic atrophy (Eye disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Herpes simplex pneumonia (Infections and infestations) | 1 | 0
Infective spondylitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Psoas abcess (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 2 | 5
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 1 | 0
Dural tear (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrong technique in device usage process (Injury, poisoning and procedural complications) | 2 | 4
Type 2 Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Mucoid degeneration of the anterior cruciate ligament (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 5
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal retrolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dorsal ramus syndrome (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 2 | 1
Spinal epidural haematoma (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 1 | 0
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0
Iliac vein perforation (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Population ANT (N=164) | Total Population POST (N=173)
Pyrexia (General disorders) | 3 (3) | 18 (19)
Procedural pain (Injury, poisoning and procedural complications) | 18 (18) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (35) | 16 (16)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (15) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT02617563/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT02617563/SAP_001.pdf